CLINICAL TRIAL: NCT05636813
Title: Usefulness of an Assistive Technology Training Program for Adolescents With Dyslexia: Pilot Study
Brief Title: Usefulness of an Assistive Technology Training Program for Adolscents With Dyslexia
Acronym: FormONC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-160
Record Dates: First submitted 2021-04-19; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-02

CONDITIONS: Dyslexia; Adolescent
Keywords: dyslexic adolescent; dyslexia; education; assistive technology
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Pilot, pronostic, open-label, non-randomized, descriptive, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): Program of training of use of assistive technology
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Patients are trained to use AT (2 sessions of 4 hours). Written langage skills, autonomy, the use are evaluated before and after training.

SUMMARY:
Specific Written Language Disorders (SWLD) are severe and lasting impairments in the development of written language that affect approximately 10% of the school-age population.Concerned patients don't have any intellectual disability.

Speech therapy help them to improve their language skills but also to compensate for their difficulties.

School environment is one of the places where these disorders can constitute a real handicap.

Given the prevalence of disorders, governments but also supra-governmental authorities have promoted educational integration of the concerned patients around the world. In France, different systems exist to help these patients with SWLD to follow an education that allows them to update their capacities as much as possible. School facilities are proposed such as attribution of Assistive Technology (AT). Nevertheless, these facilities have some limitations.

Concerning AT, several studies have shown the benefits for patients with dyslexia such as a better use of them. However, there were some limitations in their use and their usefulness.

The lack of use training is one of the barriers cited by patients and caregivers (parents and teachers).

Assistive Technology training exists for patients with dyslexia but very few studies have measured their influence on their performance in written language. Moreover, these studies did not take into account the previous level of computer practice nor the natural appropriation of the AT (ie: anyone can appropriate themselves). It is therefore difficult to affirm the specificity of the training's influence.

This study aims to assess the usefulness of AT training on the written language performance of adolescents with dyslexia. This work will study teenager's autonomy and how they use these tools.

ELIGIBILITY:
Inclusion Criteria:

* adolescents with dyslexia
* normal schooling (not in a specialized establishment)
* with attribution of assistive technology less than 3 months or planned soon or low usage

Exclusion Criteria:

* oral disabilities hindering intelligibility
* physical disabilities (hands) hindering use of AT
* auditive and visual disabilities

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reading skills without assistive technology before training: number of words read | 9 weeks
  minimum 0 and maximum 152, higher scores mean a better outcome
Reading skills without assistive technology before training: number of misread | 9 weeks
  minimum 0 and maximum 152, higher scores mean a worse outcome
Reading skills without assistive technology before training: time to read | 9 weeks
  (in seconds, higher times mean a worse outcome)
Reading comprehension skills without assistive technology before training: titles choices | 9 weeks
  (higher scores mean a better outcome, minimum 0 and maximum 6)
Reading comprehension skills without assistive technology before training: right or wrong | 9 weeks
  (higher scores mean a better outcome: minimum 0 and maximum 8)
Reading comprehension skills without assistive technology before training: choice of the good answer | 9 weeks
  (higher scores mean a better outcome:minimum 0 and maximum 4).
Reading effectiveness without assistive technology before training | 9 weeks
  sum (minimum 0 and maximum 172: higher scores mean a better outcome) of number of correct read words (minimum 0 and maximum 152) plus comprehension score (minimum 0 and maximum 18) plus reading score (0: failed, 1: partially succeded, 2 succeded)
Reading skills without assistive technology after training: number of words read | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a better outcome)
Reading skills without assistive technology after training: number of misread | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a worse outcome)
Reading skills without assistive technology after training: time to read | 9 weeks
  (in seconds, higher times mean a worse outcome)
Reading comprehension skills without assistive technology after training: titles choices | 9 weeks
  (higher scores mean a better outcome, minimum 0 and maximum 6)
Reading comprehension skills without assistive technology after training: right or wrong | 9 weeks
  (higher scores mean a better outcome: minimum 0 and maximum 8)
Reading comprehension skills without assistive technology after training: choice of the good answer | 9 weeks
  (higher scores mean a better outcome:minimum 0 and maximum 4).
Reading effectiveness without assistive technology after training | 9 weeks
  sum (minimum 0 and maximum 172: higher scores mean a better outcome) of number of correct read words (minimum 0 and maximum 152) plus comprehension score (minimum 0 and maximum 18) plus reading score (0: failed, 1: partially succeded, 2 succeded)
Reading skills with assistive technology before training: number of words read | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a better outcome)
Reading skills with assistive technology before training: number of misread | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a worse outcome)
Reading skills with assistive technology before training: time to read | 9 weeks
  (in seconds, higher times mean a worse outcome)
Reading comprehension skills with assistive technology before training: titles choices | 9 weeks
  (higher scores mean a better outcome, minimum 0 and maximum 6)
Reading comprehension skills with assistive technology before training: right or wrong | 9 weeks
  (higher scores mean a better outcome: minimum 0 and maximum 8)
Reading comprehension skills with assistive technology before training: choice of the good answer | 9 weeks
  (higher scores mean a better outcome:minimum 0 and maximum 4).
Reading effectiveness with assistive technology before training | 9 weeks
  sum (minimum 0 and maximum 172: higher scores mean a better outcome) of number of correct read words (minimum 0 and maximum 152) plus comprehension score (minimum 0 and maximum 18) plus reading score (0: failed, 1: partially succeded, 2 succeded)
Reading skills with assistive technology after training: number of words read | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a better outcome)
Reading skills with assistive technology after training: number of misread | 9 weeks
  (minimum 0 and maximum 152, higher scores mean a worse outcome)
Reading skills with assistive technology after training: time to read | 9 weeks
  (in seconds, higher times mean a worse outcome)
Reading comprehension skills with assistive technology after training: titles choices | 9 weeks
  (higher scores mean a better outcome, minimum 0 and maximum 6)
Reading comprehension skills with assistive technology after training: right or wrong | 9 weeks
  (higher scores mean a better outcome: minimum 0 and maximum 8)
Reading comprehension skills with assistive technology after training: choice of the good answer | 9 weeks
  (higher scores mean a better outcome:minimum 0 and maximum 4).
Reading effectiveness with assistive technology after training | 9 weeks
  sum (minimum 0 and maximum 172: higher scores mean a better outcome) of number of correct read words (minimum 0 and maximum 152) plus comprehension score (minimum 0 and maximum 18) plus reading score (0: failed, 1: partially succeded, 2 succeded)
Written skills without assistive technology before training | 9 weeks
  * Number of correct written words (handwriting) in 3 minutes (higher scores mean a better outcome)
  * Number of incorrect written words (handwriting) in 3 minutes (higher scores mean a worse outcome)
Written skills without assistive technology after training | 9 weeks
  * Number of correct written words (handwriting) in 3 minutes (higher scores mean a better outcome)
  * Number of incorrect written words (handwriting) in 3 minutes (higher scores mean a worse outcome)
Written skills with assistive technology before training | 9 weeks
  * Number of correct written words in 3 minutes (higher scores mean a better outcome)
  * Number of incorrect written words in 3 minutes (higher scores mean a worse outcome)
Written skills with assistive technology after training | 9 weeks
  * Number of correct written words in 3 minutes (higher scores mean a better outcome)
  * Number of incorrect written words in 3 minutes (higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Autonomy before training | 9 weeks
  Autonomy in the daily life (number of help's need) (higher scores mean a worse outcome)
Autonomy after training | 9 weeks
  Autonomy in the daily life (number of help's need) (higher scores mean a worse outcome)
Effectiveness of assistive technology utilization before training: Frequency of use | 9 weeks
  (minutes per week) (higher scores mean a better outcome)
Effectiveness of assistive technology utilization before training: Number of different utilization locations | 9 weeks
  (home, school, …) (higher scores mean a better outcome)
Effectiveness of assistive technology utilization before training: Number of different accomplished tasks | 9 weeks
  (games, homework, messaging, social networks, …) (higher scores mean a better outcome)
Effectiveness of assistive technology utilization after training: Frequency of use | 9 weeks
  (minutes per week) (higher scores mean a better outcome)
Effectiveness of assistive technology utilization after training: Number of different utilization locations | 9 weeks
  (home, school, …) (higher scores mean a better outcome)
Effectiveness of assistive technology utilization after training: Number of different accomplished tasks | 9 weeks
  (games, homework, messaging, social networks, …) (higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Desmaisons, MRS, Principal Investigator — University Hospital of Caen
Locations (1):
- Desmaisons, Caen, France